CLINICAL TRIAL: NCT02779907
Title: Prevalence and Associations of Paediatric Chronic Suppurative Otitis Media and Hearing Impairment in a Rural District of Malawi: A Cross-sectional Survey
Brief Title: Prevalence and Associations of Paediatric Chronic Suppurative Otitis Media and Hearing Impairment in Rural Malawi
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Liverpool School of Tropical Medicine (Other)
Collaborators: Kamuzu University of Health Sciences (Other); Malawi-Liverpool-Wellcome Trust Clinical Research Programme (Other)
Responsible Party: Sponsor
Other Study IDs: LOI 0182
Record Dates: First submitted 2016-05-06; First posted 2016-05-23 (Estimated); Last update posted 2016-06-06 (Estimated); Status verified 2016-06

CONDITIONS: Chronic Suppurative Otitis Media; Hearing Impairment
Keywords: Paediatric; Malawi
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study Population: Children aged 4-6 years resident in Chikwawa District.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No interventions planned for this observational study

SUMMARY:
This community-based cross-sectional survey will estimate the frequency and risk factors of Chronic Suppurative Otitis Media and Hearing Impairment in Children ages 4-6 years in the Chikwawa District. These data will be useful for service planning, disease prevention efforts and to guide future research in this field.

DETAILED DESCRIPTION:
Type of research study:

Cross sectional survey

Problem to be studied:

Chronic suppurative otitis media and hearing impairment are important causes of morbidity, affecting 4-10% of children throughout sub-Saharan Africa. Many of the causes of disease are preventable with simple interventions. There is significant variation in disease burden and causes between countries, and currently no data on the frequency and causes of disease in Malawi.

Previous studies suggest poverty, crowding, paternal smoking and indoor cooking all increase the risk of developing chronic suppurative otitis media. The associations with use of an efficient cookstove have not been studied. The causes of childhood hearing impairment vary significantly by region and include otitis, other infections and cryptogenic causes.

Objectives:

* Estimate the prevalence of CSOM and other ear pathology in a population representative sample of 4-6 year-old children in a rural district of Malawi.
* Describe associations (including household use of an efficient cookstove) of CSOM
* Estimate the prevalence of hearing impairment defined by screening audiometry in a population representative sample of 4-6 year-old children in a rural district of Malawi.
* Describe associations of hearing impairment in a population representative sample of 4-6 year-old children in a rural district of Malawi.

Methodology:

A village level cluster survey in the Chikwawa district of Malawi. The study will survey 270 children across 10 systematically determined clusters using 2008 census data. The investigators will undertake video otoscopy and basic hearing screening in the field using a validated smartphone screening tool. The research will also look for associations between chronic middle ear infection and potential risk factors for disease using negative binomial regression. This will include household use of an efficient cookstove.

Expected findings and their dissemination:

The investigators will establish the prevalence and associations of chronic suppurative otitis media and of hearing impairment in children aged 4-6 years in the Chikwawa district. The investigators hope these data will guide further development of ENT service in Malawi, and may indicate possible preventative strategies. The results will be disseminated to the communities, local health services and the College of Medicine of Malawi.

ELIGIBILITY:
Inclusion Criteria:

* Child aged 4-6 years old
* Resident in the CAPS study area in the Chikwawa district of southern Malawi
* Parental consent and child's assent to inclusion in the study

Exclusion Criteria:

* Parent/guardian of participant unable to provide informed consent to their child's participation
* Participant refusal to assent to participation
* Participant unable to explicitly assent to involvement in the study (e.g. developmental delay, learning difficulties, unwell)

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children aged 4-6 years living in the Chikwawa District
Sampling Method: Probability Sample
Enrollment: 270 (Estimated)
Dates: Start 2016-05; Primary Completion 2016-07 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Chronic Suppurative Otitis Media | Day1; This is a Cross-Sectional Survey and each participant will be assessed once. Therefore the outcome will be measured at data collection.
  Chronic Suppurative Otitis Media will be defined as per the the World Health Organisation ear and hearing survey diagnostic criteria. To assign a diagnosis, tympanic membrane images and clinical data for each participant will be reviewed by two ENT surgeons who will assign a diagnosis. Disagreements will be resolved by a third 'tiebreaker'.

SECONDARY OUTCOMES:
Hearing Impairment at more than 25 decibels hearing loss cutoff at 1000Hz, 2000Hz and 4000Hz | Day 1; This is a Cross-Sectional Survey and each participant will be assessed once. Therefore the outcome will be measured at data collection.
  Hearing impairment will be defined as per the World Health Organisation definition of mild hearing impairment (25 decibels hearing loss). Each participant's hearing will be assessed using a screening audiometer.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Mortimer, PHD, MBBS, Principal Investigator — LSTM
Locations (1):
- Malawi-Liverpool-Wellcome Trust Clinical Research Program Chikwawa District Hospital Field Research Sute, Iratu, Chikwawa, Malawi

IPD SHARING:
Plan to Share IPD: Yes
Participants will be consented for anonymised data storage for further research up to a period of 5 years following completion of the study. These data will be held on a secure server at LSTM by the principal investigator. Data may be shared with any interested parties following successful ethical review from COMREC and LSTM.